CLINICAL TRIAL: NCT00038493
Title: Phase II Evaluation Temozolomide and Farnesyl Transferase Inhibitor (SCH66336) for the Treatment of Recurrent and Progressive Glioblastoma Multiforme
Brief Title: Temozolomide and SCH66336 for Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM01-258
Record Dates: First submitted 2002-05-31; First posted 2002-06-03 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM; Glioma; Brain Tumor
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms | interventions — Temozolomide; lonafarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Temozolomide and SCH66336

SUMMARY:
This study will combine the chemotherapy agent temozolomide with the investigational drug SCH66336 (an agent which interferes with new cell growth). Patients will be treated with oral temozolomide on days 1-5 and oral SCH66336 on days 8-28 every 28 days.

DETAILED DESCRIPTION:
Temozolomide at a dose of, 150-200 mg/m2, will be administered orally, after fasting for one hour, once a day for 5 consecutive days (days 1 through 5) every 4 weeks (plus up to 3 days). The starting dose level of 200 mg/m2 will be used for patients who have not previously received any chemotherapy or at 150 mg/m2 for patients who have received previous chemotherapy.

SCH66336 will be given orally, with water, in the morning and in the evening for three weeks (Days 8 - 28) every 28 days (plus up to 3 days) 1 hour before or after morning and evening meals. Patients will take 150 mg in the morning and 150 mg in the evening.

Treatment courses may be repeated every 28 days following the first daily dose of Temozolomide for the previous course.

ELIGIBILITY:
Inclusion:

* Patients with histologically proven supratentorial glioblastoma multiforme (GBM).
* Patients must have shown unequivocal evidence for tumor recurrence or progression by MRI scan after radiation therapy. The scan done prior to study entry documenting progression will be reviewed by the primary investigator to document tumor volume changes to provide a gross assessment of growth rate.
* Patients may have had: a) no prior chemotherapy, b) 1 prior adjuvant chemotherapy, c) 1 prior adjuvant chemotherapy followed by 1 regimen for recurrent disease, or d) 1 or 2 prior chemotherapy regimens for recurrent or progressive tumor.
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of this hospital.
* Patients must have shown unequivocal evidence for tumor progression by MRI or CT scan. A scan should be performed within 14 days prior to registration and on a steroid dose that has been stable for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline MR/CT is required. The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement.
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

  1. They have recovered from the effects of surgery.
  2. Residual disease following resection of recurrent tumor is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a CT/ MRI should be done no later than 96 hours in the immediate post-operative period or at least 4 weeks post-operatively, within 14 days prior to registration. If the 96-hour scan is more than 14 days before registration, the scan needs to be repeated. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required on a stable steroid dosage for at least 5 days.
* Patients must be > 18 years old, and with life expectancy > 8 weeks.
* Patients must have a Karnofsky performance status of > 60 (Karnofsky Performance Scale; Appendix C).
* Patients must have recovered from the toxic effects of prior therapy: 4 weeks from prior cytotoxic therapy and/or at least two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.
* Patients must have adequate bone marrow function (ANC> 1,500/mm3 and platelet count of > 100,000/mm3), adequate liver function (SGPT and alkaline phosphatase <2 times normal, bilirubin <1.5 mg%), and adequate renal function (BUN and creatinine <1.5 times institutional normal) prior to starting therapy.
* Patients must have a normal QT interval on an EKG done within 2 weeks prior to study entry.
* Patients must not be taking primidone, carbamazepine, phenobarbital or phenytoin anticonvulsants. Patients changing from these anticonvulsants to others that are allowed must be off the drugs listed above for at least 72 hours.
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Patients must not have:

  1. active infection
  2. disease that will obscure toxicity or dangerously alter drug metabolism
  3. serious intercurrent medical illness.
  4. prior recurrence with either Temozolomide or a farnesyl transferase inhibitor
  5. oral contraceptives and other hormonal methods (Depo-Provera) of birth control.
* Patients must not be pregnant and both male and female patients must practice adequate contraception.

Exclusion:

* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Patients with the following are ineligible:

  1. active infection
  2. pregnancy and must practice adequate contraception
  3. disease that will obscure toxicity or dangerously alter drug metabolism
  4. serious intercurrent medical illness
  5. previous treatment with either Temozolomide or a farnesyl transferase inhibitor
  6. oral contraceptives and other hormonal methods (Depo-Provera) of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2001-09-21 (Actual); Primary Completion 2005-08-01 (Actual); Study Completion 2005-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UTMD Anderson Cancer Center, Houston, Texas, United States